CLINICAL TRIAL: NCT02676271
Title: The Long Term Outcome of Varus Derotational Osteotomy for Legg-Calvé-Perthes' Disease
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Noam Shohat, Assaf-Harofeh Medical Center
Other Study IDs: 0063-15
Record Dates: First submitted 2015-11-24; First posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Legg-Calvé-Perthes Disease
MeSH Terms: conditions — Legg-Calve-Perthes Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Procedure: Proximal varus derotational osteotomy — The purpose of surgery was to relocate the protruded, deformed femoral head from its lateral position back to the acetabulum to achieve containment. Surgery was preceded by a hip arthrography with dynamic examination to find the suitable containment position and plan the correct osteotomy angles accordingly. A sub trochanteric osteotomy was performed then after in an open or closed wedge form, with fixation in an angle that gave best coverage.
  Other Names: Femoral plate

SUMMARY:
Background: Varus derotation osteotomy (VDRO) is one of the most popular surgical treatments for Legg-Calvé-Perthes disease yet its long term results have not been assessed. Our purpose was to determine the long term clinical and radiographic outcomes of these patients.

Methods: Forty patients (43 hips) who had undergone VDRO for LCPD who participated in a long term follow-up study a decade ago were approached for the present study.

All patients were treated in our institution during 1959 to 1983 with proximal VDRO.

The patients were invited to for a medical interview and a physical examination. They were also asked to fill out questionnaires and to provide or undergo a standing anteroposterior (AP) pelvic and a lateral hip radiographs during the visit.

Patients were asked to self-grade their hip pain as none, mild, moderate or severe and to grade their back pain using the Visual Analogue Scale (VAS) between 0-10. Details regarding daily function, physical activity, work status and family history were obtained. All participants completed the Harris Hip Score (HHS) with a maximum score of 100 and the Short Form-36 which is composed of 8 sections and has a maximum score of 100.

The physical examination included an assessment of the hip range of motion, leg length discrepancy and the presence of a Trendelenburg sign.

Radiographic parameters evaluated were the Tonnis grade (with a score between 0-3), head size ratio, and the center-edge (CE) angle.

ELIGIBILITY:
Inclusion Criteria:

* All patients were treated in our institution during 1959 to 1983 with proximal VDRO and were examined a decade ago

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Forty patients (43 hips) who had undergone VDRO for LCPD who participated in a long term follow-up study a decade ago. All patients were treated in our institution during 1959 to 1983 with proximal VDRO.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes | a follow-up 42.5 years from surgery
  The hip status was assessed by the Harris Hip Score (HHS)
Clinical outcomes | a follow-up 42.5 years from surgery
  The Short Form-36 (SF-36) was used to asses the general well being
Radiographic outcomes | a follow-up 42.5 years from surgery
  The degenerative changes were assessed by The Tonnis grade.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Shohat, MD, Principal Investigator — Tel Aviv University, Israel
Locations (1):
- Assaf Haroffeh Medical center, Ẕerifin, Israel